CLINICAL TRIAL: NCT04877730
Title: Diabetes Closed-Loop Project 6 (DCLP6): Fully Automated Closed-Loop Control in Type 1 Diabetes Using Meal Anticipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sue Brown, Professor, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 210035; UC4DK108483 (NIH)
Record Dates: First submitted 2021-04-26; First posted 2021-05-07 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes (T1D); Continuous Glucose Monitor (CGM); Insulin Pump; Fully Automated Closed Loop (FCL); Hybrid Closed Loop (HCL)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- FCL (Fully Closed Loop) (Experimental): Closed-loop control without meal anticipation module without meal bolus
  Interventions: Device: Fully Closed Loop (FCL)
- FCL+ (Fully Closed Loop with meal anticipation) (Experimental): Closed-loop control with meal anticipation module without meal bolus
  Interventions: Device: Fully Closed Loop with meal anticipation module (FCL+)
- HCL (Hybrid Closed Loop) (Experimental): Closed-loop control without meal anticipation module with meal bolus
  Interventions: Device: Hybrid Closed Loop (HCL)

INTERVENTIONS:
Device: Fully Closed Loop (FCL) — Closed loop without a meal anticipation module without announced carbohydrate
  Arms: FCL (Fully Closed Loop)
Device: Fully Closed Loop with meal anticipation module (FCL+) — Closed loop with a meal anticipation module and without announced carbohydrate
  Arms: FCL+ (Fully Closed Loop with meal anticipation)
Device: Hybrid Closed Loop (HCL) — Closed loop without a meal anticipation module with announced carbohydrate
  Arms: HCL (Hybrid Closed Loop)

SUMMARY:
The purpose of this study is to test the meal anticipation module on a closed loop algorithm, assessing efficacy and safety.

DETAILED DESCRIPTION:
This is a pilot study to assess glycemic responses to three different approaches to insulin dosing for carbohydrate ingestion, with different approaches to a closed-loop system in random order;

1. without the meal anticipation module and without carbohydrate announcement (FCL)
2. with the meal anticipation module and without carbohydrate announcement (FCL+)
3. without the meal anticipation module and with carbohydrate announcement (HCL),

This study will target completion of up to 36 adults in a randomized cross-over trial, comparing blood glucose time in range 70-180 mg/dL following meals with and without the meal anticipation module in use (FCL+ vs FCL), and comparing to a system with carb announcement instead of a meal anticipation module (HCL). The study will also assess safety when dinner is consumed later than usual and when a lunch is consumed without having been entrained in the meal anticipation module. Each participant will complete each of the 3 modules in random order.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18.0 and ≤70 years old at time of consent
2. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year
3. Currently using insulin for at least six months
4. Currently using insulin pump for at least three months
5. Using insulin parameters such as carbohydrate ratio and correction factors consistently on their pump in order to dose insulin for meals or corrections
6. Access to internet and willingness to upload data during the study as needed
7. For females, not currently known to be pregnant or breastfeeding
8. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of childbearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
9. Willingness to suspend use of any personal CGM for the duration of the clinical trial once the study CGM is in use
10. Willingness to use the University of Virginia (UVa) closed-loop system throughout study admission
11. Willingness to use the insulin supplied by the study for the hotel stay, if not already using that preparation. Study insulin will be lispro (Humalog) or aspart (Novolog)
12. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial (including metformin, GLP-1 agonists, pramlintide, DPP-4 inhibitors, biguanides, sulfonylureas and naturaceuticals)
13. Willingness to eat at least 1g/kg of carbohydrate per day during the hotel admission
14. Willingness to reschedule if placed on oral steroids
15. An understanding and willingness to follow the protocol and signed informed consent
16. Willingness to commit to self-quarantine for at least 5 days before COVID-19 testing (If participant has received a full course of COVID-19 vaccine and data emerge suggesting significantly reduced transmissibility among those receiving that vaccine, this self-quarantine requirement can be waived.)

Exclusion Criteria:

1. History of diabetic ketoacidosis (DKA) in the 12 months prior to enrollment
2. Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment
3. Pregnancy or intent to become pregnant during the trial
4. Currently being treated for a seizure disorder
5. Planned surgery during study duration
6. Treatment with any non-insulin glucose-lowering agent (including metformin, GLP-1 agonists, pramlintide, DPP-4 inhibitors, SGLT-2 inhibitors, biguanides, sulfonylureas and naturaceuticals)
7. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol.
8. Use of an automated insulin delivery mechanism that is not downloadable by the subject or study team
9. Known contact with a COVID-19 positive individual within 14 days of the hotel/rental house studies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Brown, MD, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH Data Sharing Policy and Implementation Guidance on sharing research resources for research purposes to qualified individuals within the scientific community.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Generally data will be made available after the primary publications of each study.
Access Criteria: Data Sharing agreements will be formulated by the study team.

REFERENCES:
- [Result] Garcia-Tirado J, Colmegna P, Villard O, Diaz JL, Esquivel-Zuniga R, Koravi CLK, Barnett CL, Oliveri MC, Fuller M, Brown SA, DeBoer MD, Breton MD. Assessment of Meal Anticipation for Improving Fully Automated Insulin Delivery in Adults With Type 1 Diabetes. Diabetes Care. 2023 Sep 1;46(9):1652-1658. doi: 10.2337/dc23-0119. PMID 37478323

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 50 participants signed informed consent between May 2021 and March 2022. Four did not pass screening and ten participants withdrew prior to randomization. Thirty-six were randomized and the trial was completed by 35 (97%) participants; one participant was excluded after randomization.
Pre-assignment Details: A minimum of 14 days of CGM and pump information were required for analysis of baseline glycemic control, meal patterns, and insulin use. For participants already using a Dexcom G6, retrospective data prior to enrollment could be used. Participants not using a Dexcom G6 CGM were trained and sent equipment for a minimum 30 days of data prior to study admission. Participants were asked to keep daily meal records to determine the "expected" timing of breakfast and dinner for the admission.
Groups:
- Fully Closed Loop (FCL) , Fully Closed Loop With Meal Anticipation (FCL+), Hybrid Closed Loop (HCL): Participants completed three 24 hour sequential assessments of the closed loop control modalities in randomized order in a supervised hotel environment. At the end of each 24-hour period participants were transferred to the next controller modalities following the randomization order.
  The three 24-hour study periods were designed to be as similar as possible with respect to the timing and content of food and activity. On each day, participants ate dinner 1.5 hours after the "expected" time from the Baseline analysis and ate breakfast at the "expected" time. Lunch was at 13:00. On the HCL day, participants informed the control system of the carbohydrates they intended to eat prior to the meal. On FCL and FCL+ days, no manual bolus was given at mealtimes. A mid-afternoon snack of carbohydrate-free food (deli meat and/or cheese) was provided at 4 pm if desired (and repeated every day if taken).
  At 10:30 a.m. for each study period, participants together went on a light walk for 25 minutes.
  Participants in this group completed the three 24 hour admissions in the following order: FCL, FCL+, HCL.
  Fully Closed Loop (FCL): Closed-loop control without meal anticipation module without meal bolus. Fully Closed Loop with meal anticipation module (FCL+): Closed-loop control with meal anticipation module without meal bolus. Hybrid Closed Loop (HCL): Closed-loop control without meal anticipation module with meal bolus.
- FCL (Fully Closed Loop), HCL (Hybrid Closed Loop), FCL+ (Fully Closed Loop With Meal Anticipation): Participants completed three 24 hour sequential assessments of the closed loop control modalities in randomized order in a supervised hotel environment. At the end of each 24-hour period participants were transferred to the next controller modalities following the randomization order.
  The three 24-hour study periods were designed to be as similar as possible with respect to the timing and content of food and activity. On each day, participants ate dinner 1.5 hours after the "expected" time from the Baseline analysis and ate breakfast at the "expected" time. Lunch was at 13:00. On the HCL day, participants informed the control system of the carbohydrates they intended to eat prior to the meal. On FCL and FCL+ days, no manual bolus was given at mealtimes. A mid-afternoon snack of carbohydrate-free food (deli meat and/or cheese) was provided at 4 pm if desired (and repeated every day if taken).
  At 10:30 a.m. for each study period, participants together went on a light walk for 25 minutes.
  Participants in this group completed the three 24 hour admissions in the following order: FCL, HCL, FCL+.
  Fully Closed Loop (FCL): Closed-loop control without meal anticipation module without meal bolus. Hybrid Closed Loop (HCL): Closed-loop control without meal anticipation module with meal bolus. Fully Closed Loop with meal anticipation module (FCL+): Closed-loop control with meal anticipation module without meal bolus.
- FCL+ (Fully Closed Loop With Meal Anticipation), FCL (Fully Closed Loop), HCL (Hybrid Closed Loop): Participants completed three 24 hour sequential assessments of the closed loop control modalities in randomized order in a supervised hotel environment. At the end of each 24-hour period participants were transferred to the next controller modalities following the randomization order.
  The three 24-hour study periods were designed to be as similar as possible with respect to the timing and content of food and activity. On each day, participants ate dinner 1.5 hours after the "expected" time from the Baseline analysis and ate breakfast at the "expected" time. Lunch was at 13:00. On the HCL day, participants informed the control system of the carbohydrates they intended to eat prior to the meal. On FCL and FCL+ days, no manual bolus was given at mealtimes. A mid-afternoon snack of carbohydrate-free food (deli meat and/or cheese) was provided at 4 pm if desired (and repeated every day if taken).
  At 10:30 a.m. for each study period, participants together went on a light walk for 25 minutes.
  Participants in this group completed the three 24 hour admissions in the following order: FCL+, FCL, HCL.
  Fully Closed Loop with meal anticipation module (FCL+): Closed-loop control with meal anticipation module without meal bolus. Fully Closed Loop (FCL): Closed-loop control without meal anticipation module without meal bolus. Hybrid Closed Loop (HCL): Closed-loop control without meal anticipation module with meal bolus.
- FCL+ (Fully Closed Loop With Meal Anticipation), HCL(Hybrid Closed Loop), FCL(Fully Closed Loop): Participants completed three 24 hour sequential assessments of the closed loop control modalities in randomized order in a supervised hotel environment. At the end of each 24-hour period participants were transferred to the next controller modalities following the randomization order.
  The three 24-hour study periods were designed to be as similar as possible with respect to the timing and content of food and activity. On each day, participants ate dinner 1.5 hours after the "expected" time from the Baseline analysis and ate breakfast at the "expected" time. Lunch was at 13:00. On the HCL day, participants informed the control system of the carbohydrates they intended to eat prior to the meal. On FCL and FCL+ days, no manual bolus was given at mealtimes. A mid-afternoon snack of carbohydrate-free food (deli meat and/or cheese) was provided at 4 pm if desired (and repeated every day if taken).
  At 10:30 a.m. for each study period, participants together went on a light walk for 25 minutes.
  Participants in this group completed the three 24 hour admissions in the following order: FCL+, HCL, FCL.
  Fully Closed Loop with meal anticipation module (FCL+): Closed-loop control with meal anticipation module without meal bolus. Hybrid Closed Loop (HCL): Closed-loop control without meal anticipation module with meal bolus. Fully Closed Loop (FCL): Closed-loop control without meal anticipation module without meal bolus.
- HCL (Hybrid Closed Loop), FCL (Fully Closed Loop), FCL+ (Fully Closed Loop With Meal Anticipation): Participants completed three 24 hour sequential assessments of the closed loop control modalities in randomized order in a supervised hotel environment. At the end of each 24-hour period participants were transferred to the next controller modalities following the randomization order.
  The three 24-hour study periods were designed to be as similar as possible with respect to the timing and content of food and activity. On each day, participants ate dinner 1.5 hours after the "expected" time from the Baseline analysis and ate breakfast at the "expected" time. Lunch was at 13:00. On the HCL day, participants informed the control system of the carbohydrates they intended to eat prior to the meal. On FCL and FCL+ days, no manual bolus was given at mealtimes. A mid-afternoon snack of carbohydrate-free food (deli meat and/or cheese) was provided at 4 pm if desired (and repeated every day if taken).
  At 10:30 a.m. for each study period, participants together went on a light walk for 25 minutes.
  Participants in this group completed the three 24 hour admissions in the following order: HCL, FCL, FCL+.
  Hybrid Closed Loop (HCL): Closed-loop control without meal anticipation module with meal bolus. Fully Closed Loop (FCL): Closed-loop control without meal anticipation module without meal bolus. Fully Closed Loop with meal anticipation module (FCL+): Closed-loop control with meal anticipation module without meal bolus.
- HCL (Hybrid Closed Loop), FCL+ (Fully Closed Loop With Meal Anticipation), FCL(Fully Closed Loop): Participants completed three 24 hour sequential assessments of the closed loop control modalities in randomized order in a supervised hotel environment. At the end of each 24-hour period participants were transferred to the next controller modalities following the randomization order.
  The three 24-hour study periods were designed to be as similar as possible with respect to the timing and content of food and activity. On each day, participants ate dinner 1.5 hours after the "expected" time from the Baseline analysis and ate breakfast at the "expected" time. Lunch was at 13:00. On the HCL day, participants informed the control system of the carbohydrates they intended to eat prior to the meal. On FCL and FCL+ days, no manual bolus was given at mealtimes. A mid-afternoon snack of carbohydrate-free food (deli meat and/or cheese) was provided at 4 pm if desired (and repeated every day if taken).
  At 10:30 a.m. for each study period, participants together went on a light walk for 25 minutes.
  Participants in this group completed the three 24 hour admissions in the following order: HCL, FCL+, FCL.
  Hybrid Closed Loop (HCL): Closed-loop control without meal anticipation module with meal bolus. Fully Closed Loop with meal anticipation module (FCL+): Closed-loop control with meal anticipation module without meal bolus. Fully Closed Loop (FCL): Closed-loop control without meal anticipation module without meal bolus.
Period: Overall Study
Arm/Group | Fully Closed Loop (FCL) , Fully Closed Loop With Meal Anticipation (FCL+), Hybrid Closed Loop (HCL) | FCL (Fully Closed Loop), HCL (Hybrid Closed Loop), FCL+ (Fully Closed Loop With Meal Anticipation) | FCL+ (Fully Closed Loop With Meal Anticipation), FCL (Fully Closed Loop), HCL (Hybrid Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation), HCL(Hybrid Closed Loop), FCL(Fully Closed Loop) | HCL (Hybrid Closed Loop), FCL (Fully Closed Loop), FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop), FCL+ (Fully Closed Loop With Meal Anticipation), FCL(Fully Closed Loop)
Started | 5 | 7 | 7 | 8 | 4 | 5
Completed | 5 | 6 | 7 | 8 | 4 | 5
Not Completed | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of all study participants regardless of randomization.
Groups:
- All Participants: Baseline characteristics of all study participants regardless of randomization.
Arm/Group | All Participants
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 32
  More than one race | 0
  Unknown or Not Reported | 1
HbA1c [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] — HbA1c is measured here as a percentage instead of mmol/mol.
  percentage of glycated hemoglobin | 6.7 (0.9)
Diabetes duration (years) [Mean (Standard Deviation); unit: years] — A measure in years of how long participants have had Type 1 Diabetes.
  years | 26 (14)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.6 (5.3)
Previous CGM users [Count of Participants; unit: Participants] | 34

OUTCOME MEASURES:

1. Primary Outcome: Time in Range (TIR) 70-180 mg/dL From Breakfast Time + 5 Hours
Description: Frequency of CGM values falling between 70 mg/dL and 180mg/dL (included) in the 5 hours following breakfast. Higher TIR is a positive outcome.
Time Frame: The 5 hour period following breakfast during the study admission
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 58 (21) | 63 (19) | 75 (23)

2. Secondary Outcome: Time in Range (TIR) 70-180 mg/dL Overall
Description: Frequency of CGM values falling between 70 mg/dL and 180mg/dL (included) during the 24hr study admission. Higher TIR is a positive outcome.
Time Frame: The 24 hour study admission from 4pm to 4pm
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 77 (11) | 77 (12) | 86 (10)

3. Secondary Outcome: Time in Range (TIR) 70-180 mg/dL From Dinner Time + 5 Hours
Description: Frequency of CGM values falling between 70 mg/dL and 180mg/dL (included) in the 5 hours following dinner. Higher TIR is a positive outcome.
Time Frame: The 5 hour period following dinner during the study admission
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 72 (29) | 71 (34) | 88 (20)

4. Secondary Outcome: Time in Range (TIR) 70-180 mg/dL From Lunch Time + 5 Hours
Description: Frequency of CGM values falling between 70 mg/dL and 180mg/dL (included) in the 5 hours following lunch. Higher TIR is a positive outcome.
Time Frame: The 5 hour period following lunch during the study admission
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 65 (28) | 61 (29) | 84 (22)

5. Secondary Outcome: Time Below Range (TBR) From Breakfast Time + 5 Hours
Description: Frequency of CGM values falling below 70 mg/dL (excluded) in the 5 hours following breakfast.
Time Frame: The 5 hour period following breakfast during the study admission
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 0 [0 to 4.4] | 0 [0 to 0] | 0 [0 to 1.6]

6. Secondary Outcome: Time Below Range (TBR) Overall
Description: Frequency of CGM values falling below 70 mg/dL (excluded) during the 24hr study admission.
Time Frame: The 24 hour study admission from 4pm to 4pm
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 1.4 [0 to 4.5] | 0.3 [0 to 1.9] | 1.0 [0 to 3.5]

7. Secondary Outcome: Time Below Range (TBR) From Dinner Time + 5 Hours
Description: Frequency of CGM values falling below 70 mg/dL (excluded) in the 5 hours following dinner.
Time Frame: The 5 hour period following dinner during the study admission
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 0 [0 to 0.8] | 0 [0 to 0] | 0 [0 to 1.7]

8. Secondary Outcome: Time Below Range (TBR) From Lunch Time + 5 Hours
Description: Frequency of CGM values falling below 70 mg/dL (excluded) in the 5 hours following lunch.
Time Frame: The 5 hour period following lunch during the study admission
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

9. Secondary Outcome: Time Above Range (TAR) From Breakfast Time + 5 Hours
Description: Frequency of CGM values falling above 180 mg/dL (excluded) in the 5 hours following breakfast.
Time Frame: The 5 hour period following breakfast during the study admission
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 39 (21) | 34 (20) | 22 (24)

10. Secondary Outcome: Time Above Range (TAR) Overall
Description: Frequency of CGM values falling above 180 mg/dL (excluded) during the 24hr study admission.
Time Frame: The 24 hour study admission from 4pm to 4pm
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 20 (11) | 21 (12) | 12 (10)

11. Secondary Outcome: Time Above Range (TAR) From Dinner Time + 5 Hours
Description: Frequency of CGM values falling above 180 mg/dL (excluded) in the 5 hours following dinner.
Time Frame: The 5 hour period following dinner during the study admission
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 26 (29) | 29 (34) | 9.6 (20)

12. Secondary Outcome: Time Above Range (TAR) From Lunch Time + 5 Hours
Description: Frequency of CGM values falling above 180 mg/dL (excluded) in the 5 hours following lunch.
Time Frame: The 5 hour period following lunch during the study admission
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 33 (28) | 38 (29) | 15 (21)

13. Secondary Outcome: Time in Significant Hyperglycemia From Breakfast Time + 5 Hours
Description: Frequency of CGM values falling above 250 mg/dL (excluded) in the 5 hours following breakfast.
Time Frame: The 5 hour period following breakfast during the study admission
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 0 [0 to 9.5] | 0 [0 to 1.9] | 0 [0 to 0]

14. Secondary Outcome: Time in Significant Hyperglycemia Overall
Description: Frequency of CGM values falling above 250 mg/dL (excluded) during the 24hr study admission.
Time Frame: The 24 hour study admission from 4pm to 4pm
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 1 [0 to 4.2] | 0 [0 to 5.6] | 0 [0 to 3.5]

15. Secondary Outcome: Time in Significant Hyperglycemia From Dinner Time + 5 Hours
Description: Frequency of CGM values falling above 250 mg/dL (excluded) in the 5 hours following dinner.
Time Frame: The 5 hour period following dinner during the study admission
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

16. Secondary Outcome: Time in Significant Hyperglycemia From Lunch Time + 5 Hours
Description: Frequency of CGM values falling above 250 mg/dL (excluded) in the 5 hours following lunch.
Time Frame: The 5 hour period following lunch during the study admission
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 0 [0 to 1.82] | 0 [0 to 14.64] | 0 [0 to 0]

17. Secondary Outcome: Time in Significant Hypoglycemia From Breakfast Time +5 Hours
Description: Frequency of CGM values falling below 54 mg/dL (excluded) in the 5 hours following breakfast.
Time Frame: The 5 hour period following breakfast during the study admission
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

18. Secondary Outcome: Time in Significant Hypoglycemia Overall
Description: Frequency of CGM values falling below 54 mg/dL (excluded) during the 24hr study admission.
Time Frame: The 24 hour study admission from 4pm to 4pm
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

19. Secondary Outcome: Time in Significant Hypoglycemia Dinner Time + 5 Hours
Description: Frequency of CGM values falling below 54 mg/dL (excluded) in the 5 hours following dinner.
Time Frame: The 5 hour period following dinner during the study admission
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

20. Secondary Outcome: Time in Significant Hypoglycemia Lunch Time + 5 Hours
Description: Frequency of CGM values falling below 54 mg/dL (excluded) in the 5 hours following lunch
Time Frame: The 5 hour period following lunch during the study admission
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
percentage of time | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

21. Secondary Outcome: Number of Hypoglycemia Events From Breakfast Time + 5 Hours
Description: Number of hypoglycemia events in the 5 hours following breakfast. A hypoglycemia event is defined as at least two consecutive CGM values <70mg/dL or a hypoglycemia treatment (two events separated by less than 30 minutes are counted as one). Metrics are number of hypoglycemia events per participant.
Time Frame: The 5 hour period following breakfast during the study admission
Measure: Median (Inter-Quartile Range); unit: events per participant
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
events per participant | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

22. Secondary Outcome: Number of Hypoglycemia Events Overall
Description: Number of hypoglycemia events during the 24hr study admission. A hypoglycemia event is defined as at least two consecutive CGM values <70mg/dL or a hypoglycemia treatment (two events separated by less than 30 minutes are counted as one). Values reported as the number of hypoglycemia events per participant.
Time Frame: The 24 hour study admission from 4pm to 4pm
Measure: Median (Inter-Quartile Range); unit: events per participant
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
events per participant | 0 [0 to 1.5] | 0 [0 to 1] | 0 [0 to 2]

23. Secondary Outcome: Number of Hypoglycemia Events Dinner Time + 5 Hours
Description: Number of hypoglycemia events in the 5 hours following dinner. A hypoglycemia event is defined as at least two consecutive CGM values <70mg/dL or a hypoglycemia treatment (two events separated by less than 30 minutes are counted as one). Values reported as the number of hypoglycemia events per participant.
Time Frame: The 5 hour period following dinner during the study admission
Measure: Median (Inter-Quartile Range); unit: events per participant
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
events per participant | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

24. Secondary Outcome: Number of Hypoglycemia Events Lunch Time + 5 Hours
Description: Number of hypoglycemia events in the 5 hours following lunch. A hypoglycemia event is defined as at least two consecutive CGM values <70mg/dL or a hypoglycemia treatment (two events separated by less than 30 minutes are counted as one).
Time Frame: The 5 hour period following lunch during the study admission
Measure: Median (Inter-Quartile Range); unit: events per participant
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
events per participant | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

25. Secondary Outcome: Units of Insulin Injected Between 2 Hours Before and 5 Hours After Breakfast
Description: Sum of all system provided insulin for breakfast (as planned) post-prandial excursion, including anticipation
Time Frame: The 7 hour period including the two hours before and the 5 hours after breakfast
Measure: Mean (Standard Deviation); unit: units of insulin / kg
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
units of insulin / kg | 0.14 (0.05) | 0.14 (0.06) | 0.18 (0.10)

26. Secondary Outcome: Units of Insulin Injected (Units/kg) Overall
Description: Calculation of all system-provided insulin (units/kg) injected during the 24hr study admission.
Time Frame: The 24 hour study admission from 4pm to 4pm
Measure: Mean (Standard Deviation); unit: units of insulin / kg
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
units of insulin / kg | 0.5 (0.2) | 0.5 (0.2) | 0.6 (0.25)

27. Secondary Outcome: Units of Insulin Injected Between 2 Hours Before and 5 Hours After Dinner
Description: Sum of all system provided insulin for dinner (late) post-prandial excursion, including anticipation
Time Frame: The 7 hour period including the 2 hours before and 5 hours after dinner
Measure: Mean (Standard Deviation); unit: units of insulin / kg
Arm/Group | FCL (Fully Closed Loop) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
Number analyzed (Participants) | 35 | 35 | 35
units of insulin / kg | 0.02 (0.03) | 0.03 (0.02) | 0.02 (0.02)

ADVERSE EVENTS:
Time Frame: The AE data were reported in randomized participants for the remaining duration of their participation in the trial (up to approximately 2 weeks from randomization). 1 participant was randomized and started the trial in FCL phase but was withdrawn due to an AE and did not start the FCL+ or HCL phase.
Groups:
- Fully Closed Loop (FCL): Fully Closed Loop (FCL): Closed-loop control without meal anticipation module without meal bolus. Fully Closed Loop with meal anticipation module.
- FCL+ (Fully Closed Loop With Meal Anticipation): (FCL+): Closed-loop control with meal anticipation module without meal bolus.
- HCL (Hybrid Closed Loop): Hybrid Closed Loop (HCL): Closed-loop control without meal anticipation module with meal bolus.
Arm/Group | Fully Closed Loop (FCL) | FCL+ (Fully Closed Loop With Meal Anticipation) | HCL (Hybrid Closed Loop)
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 1/36 | 0/35 | 1/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fully Closed Loop (FCL) (N=36) | FCL+ (Fully Closed Loop With Meal Anticipation) (N=35) | HCL (Hybrid Closed Loop) (N=35)
Persistent hyperglycemia and ketonemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) — One case of persistent hyperglycemia and ketonemia that required multiple site changes and manual insulin dosing by the study team from the time of study admission (this participant was discharged from the study and data was not used).
Emesis followed by ketonemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — A case of emesis followed by ketonemia from unclear etiology but suspected gastroenteritis that occurred just prior to study completion (these final two hours of data were excluded from the analysis).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT04877730/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT04877730/ICF_001.pdf